CLINICAL TRIAL: NCT05781997
Title: Prevalence of Refractive Errors in Primary School Children in The New Valley
Brief Title: Prevalence of Refractive Errors in Primary School Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Anwar Mohamed Said, Mut ,The New Valley , Egypt, Assiut University
Other Study IDs: refractive errors
Record Dates: First submitted 2023-03-05; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cycloplegic refraction — Cycloplegic autorefraction will be attempted on all children using a table-mounted autorefractor . Cycloplegia will be achieved with three drops of 1% cyclopentolate administered 5 min apart and autorefractive measurements will be performed 30 min after the instillation of the last drop. Auto refraction readings of three consecutive measurements will be obtained and the average will be computed automatically in each eye. Each child will be reexamined until three measurements fell within 0.50 diopters (D) if any two measurements varied by >0.50D.

SUMMARY:
The study aim to determine the prevalence of refractive errors in primary school children aged 6-12 in The New Valley , Egypt .

DETAILED DESCRIPTION:
The refractive state of the eye changes as the eye's axial length increases and the cornea and lens flattens. In general, eyes are hyperopic at birth, and become slightly more hyperopic until the age of 7, at this point we see a myopic shift toward Plano until the eyes reach their adult dimensions, usually by about the age of 16.

ELIGIBILITY:
Inclusion Criteria:

Age: 6 -12-year-old Myopia :- 0.5 D to -10D Hypermetropia: 1 D to 8 D Astigmatism: 0 to 6 D Distance correction: 0.1 logs MAR (20/25 ) or better

Exclusion Criteria:

Retinopathy, Prematurity, history of genetic disease, connective tissue diseases (e.g. Stickler or Marfan syndromes, any ocular diseases, Glaucoma, Cataract, Squint.

Ages: 6 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Primary school children aged 6-12 in New Valley, Egypt not complaining from any diseases .
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
prevalence of refractive error in primary school children | baseline
  determine the prevalence of refractive error in primary school children aged 6-12 in New Valley, Egypt .

SECONDARY OUTCOMES:
Degree of Visual aquity improvement of children. | Baseline
  We need to measure : 1-Degree of improvement of visual aquity among those children .
  2 - Acceptence of the parents and children to wear spectecles among those population .

CONTACTS AND LOCATIONS:
Overall Officials: Omar Mo Ali, Professor, Study Director — supervisor; Ahmed Mh fahmy, AssProfessor, Study Director — supervisor; Mohammed An Sayed, Lecturer, Study Director — supervisor; Doaa An Mohammed, Resident, Principal Investigator — Investigator

REFERENCES:
- [Background] Donahue SP. Prescribing spectacles in children: a pediatric ophthalmologist's approach. Optom Vis Sci. 2007 Feb;84(2):110-4. doi: 10.1097/OPX.0b013e318031b09b. PMID 17299340
- [Background] Glascoe FP. Parents' evaluation of developmental status: how well do parents' concerns identify children with behavioral and emotional problems? Clin Pediatr (Phila). 2003 Mar;42(2):133-8. doi: 10.1177/000992280304200206. PMID 12659386
- [Background] Friedman DS, Repka MX, Katz J, Giordano L, Ibironke J, Hawes P, Burkom D, Tielsch JM. Prevalence of decreased visual acuity among preschool-aged children in an American urban population: the Baltimore Pediatric Eye Disease Study, methods, and results. Ophthalmology. 2008 Oct;115(10):1786-95, 1795.e1-4. doi: 10.1016/j.ophtha.2008.04.006. Epub 2008 Jun 5. PMID 18538407
- See also: Distribution of refractive error among chinese primary school children in a rural area in Pahang, Malaysia — https://pubmed.ncbi.nlm.nih.gov/35440969/